CLINICAL TRIAL: NCT02662192
Title: Targeting Functional Fitness, Hearing and Health-Related Quality of Life in Older Adults With Hearing Loss. Walk, Talk and Listen for Your Life, A Randomized Controlled Trial
Brief Title: Fitness, Hearing and Quality of Life in Older Adults With Hearing Loss. Walk, Talk and Listen for Your Life
Acronym: WTL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Charlotte Jones, Associate Professor of Medicine, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H15-02319
Record Dates: First submitted 2016-01-14; First posted 2016-01-25 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Hearing Loss, Functional
MeSH Terms: conditions — Hearing Loss, Functional | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Exercise + health education + auditory rehabilitation 10 weeks of exercise, interactive health education, socialization and auditory rehabilitation program
  Interventions: Other: Exercise + health education+ auditory rehabilitation
- Auditory rehabilitation alone (Active Comparator): auditory rehabilitation alone
  1 hour of group auditory rehabilitation once a week for 10 weeks
  Interventions: Other: auditory rehabilitation alone

INTERVENTIONS:
Other: Exercise + health education+ auditory rehabilitation — comparison of 3/4 of an hour balance, resistance and strength training, 1 hour health education, 1 hour auditory rehabilitation
  Arms: Intervention
Other: auditory rehabilitation alone — 10 weeks of one hour per week of group auditory rehabilitation
  Arms: Auditory rehabilitation alone

SUMMARY:
This study examines the effect of an exercise and health education/auditory rehabilitation and socialization intervention on functional fitness, hearing handicap and psychosocial distress measures in older adults with hearing loss.

DETAILED DESCRIPTION:
Hearing loss is associated with functional fitness declines and increased risk for isolation, dementia, depression, falls, hospitalization and premature mortality. No studies have determined the effect of an exercise intervention on these measures in older adults with hearing loss.

After baseline assessment of function fitness and several psychosocial measures, 60 older adults with hearing loss will be randomized into a 10 week exercise, health education, socialization and auditory rehabilitation program or auditory rehabilitation alone. The exercise program consists of 3/4 of an hour strengthening and resistance training followed by 30 minutes of group walking. The educational session content is determined by participants and is interactive and may include such topics as wills and probate, diabetes treatment, healthy exercise etc. The 3/4 of an hour auditory rehabilitation sessions are modified from an online program and will include interactive sessions on education about hearing and hearing devices/technologies, psychosocial support and enhancing communication skills.

At the end of the 10 week intervention the assessments of functional fitness and psychosocial measures will be repeated. The group that was randomized to the auditory rehabilitation alone will then be offered the exercise program.

ELIGIBILITY:
Inclusion criteria:

-Gender: Male and female

Age limits:

* Minimum age: 65 years of age
* Maximum age: 90 years of age.
* Self-reported diagnosis of hearing loss
* Must be independently ambulatory (no use of cane, walker or wheelchair)
* Less than150 minutes per week of self-reported physical activity
* Healthy enough to participate in the intervention without exacerbating any existing symptomatology
* Not having participated in any organized exercise program for at least 6 months
* Availability and willingness to attend at least 80% of the 10 week intervention sessions in addition to baseline and final assessments. -Be English speaking and able to sign written informed consent
* A Hearing Handicap In the Elderly-25 questionnaire score of 25 > 17

Exclusion Criteria:

* Dementia
* Depression

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
functional fitness | 3 months
  Gait speed (6 minute walk test: distance in meters walked in 6 minutes)

SECONDARY OUTCOMES:
Psychosocial outcomes | 3 months
  Hearing and health-related quality of life HHIE-25
Physical and behaviour measures | 3 months
  Physical activity: Time spent in moderate-vigorous physical activity: The Actigraph GT3X+ tri-axial waist worn accelerometer (Actigraph, Pensacola, Florida)
Project evaluation | 3 months
  Satisfaction with the Auditory Rehabilitation, health education and exercise sessions. Confidence in being able to maintain their newly acquired communication strategies and exercise regime. Comments on how the program could be improved.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Jones, PhD, MD, Principal Investigator — University of British Columbia Okanagan, Kelowna, British Columbia, Canada
Locations (1):
- Southern Medical Program, University of British Columbia Okanagan, 321 Reichwald Health Sciences Center, 1088 Discovery Ave., Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared. Consent form indicates this as well, so participants understand that their individual data will not be shared

REFERENCES:
- [Background] Jones CA, Siever J, Knuff K, Van Bergen C, Mick P, Little J, Jones G, Murphy MA, Kurtz D, Miller H. Walk, Talk and Listen: a pilot randomised controlled trial targeting functional fitness and loneliness in older adults with hearing loss. BMJ Open. 2019 Apr 14;9(4):e026169. doi: 10.1136/bmjopen-2018-026169. PMID 30987987
- [Derived] Lambert J, Ghadry-Tavi R, Knuff K, Jutras M, Siever J, Mick P, Roque C, Jones G, Little J, Miller H, Van Bergen C, Kurtz D, Murphy MA, Jones CA. Targeting functional fitness, hearing and health-related quality of life in older adults with hearing loss: Walk, Talk 'n' Listen, study protocol for a pilot randomized controlled trial. Trials. 2017 Jan 28;18(1):47. doi: 10.1186/s13063-017-1792-z. PMID 28129779

DOCUMENTS (2):
  • Informed Consent Form (2016-02-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT02662192/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-10-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT02662192/Prot_SAP_001.pdf